CLINICAL TRIAL: NCT03905733
Title: The Effects of High-flow Nasal Oxygen on Oxygenation During Rigid Bronchoscopy Under General Anesthesia in Pediatric Patients: A Prospective Observational Pilot Study
Brief Title: The Effects of High-flow Nasal Oxygen on Oxygenation During Rigid Bronchoscopy Under General Anesthesia in Pediatric Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2019-0009
Record Dates: First submitted 2019-04-02; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Foreign Bodies; Tumor; Stenosis of Trachea; Bronchus
MeSH Terms: conditions — Foreign Bodies; Neoplasms; Tracheal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- general anesthesia with rigid bronchoscopy: Patients 7 years or younger who undergo general anesthesia with rigid bronchoscopy
  Interventions: Device: Optiflow

INTERVENTIONS:
Device: Optiflow — supply of oxygen at 2 L / min/ kg through Optiflow

SUMMARY:
The aim of this study is to evaluate the effect of high-flow nasal cannula oxygen administration on maintenance of oxygenation and removal of carbon dioxide during apnoeic period in pediatric patients undergoing general anesthesia with rigid bronchoscopy

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients undergoing general anesthesia with stent placement or bougination, biopsy or removal of a foreign body or a mass through a rigid bronchoscope
* 2. Patients aged 7 or younger who meet American Society of Anesthesiologists (ASA) physical class 2-4

Exclusion Criteria:

* 1. Patients undergoing extracorporeal membrane oxygenation (ECMO)
* 2. Patients with active nasal bleeding), severe nasal obstruction, recent nasal trauma of surgery
* 3. Patients with current maxillofacial trauma or basal skull fracture
* 4. Patients with active nasal bleeding), severe nasal obstruction, recent nasal trauma of surgery
* 5. Extremely low birth weight infant and premature infant less than 28 weeks gestation age
* 6. Patients who had previously undergone rigid bronchoscopy / surgery
* 7. If the parent of subject includes a person who can not read the written consent (eg, illiterate, foreigner, etc.)

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients 7 years or younger who undergo general anesthesia with rigid bronchoscopy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Hypoxia occurs the first time | The time taken to reach the point at which peripheral oxygen saturation fell below 90% for the first time immediately after the onset of apnea intraoperatively.
  The time taken to reach the point at which peripheral oxygen saturation fell below 90 for the first time immediately after the onset of apnea
the lowest oxygen saturation | apnea period during the rigidbroscopic procedure/surgery
  the lowest value of oxygen saturation measured percutaneously at extremity.
Occurence of hypoxic event | apnea period during the rigidbroscopic procedure/surgery
  Occurence of hypoxic event: Presence or absence of hypoxia(peripheral oxygen saturation fell below 90% ) during rigid bronchoscopy

SECONDARY OUTCOMES:
End-tidal carbon dioxide partial pressure | end-tidal CO2 partial pressure after 3 consecutive breaths after intubation or insertion of laryngeal mask following end of apnea during intraoperative period.
Arterial oxygen / carbon dioxide partial pressure | shortly before start of apnea (within 30 seconds) and shortly after end of apnea (within 30 seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic and Cardiovascular Surgery, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided